CLINICAL TRIAL: NCT04062734
Title: Endovascular Treatment of Aorto-iliac Disease Using in Situ Fenestration
Acronym: PREFISIT
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190689
Record Dates: First submitted 2019-07-01; First posted 2019-08-20 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2020-12

CONDITIONS: Peripheral Artery Disease; Abdominal Aortic Aneurysm
Keywords: Peripheral artery disease; abdominal aortic aneurysm; in situ fenestration; endovascular treatment
MeSH Terms: conditions — Peripheral Arterial Disease; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In situ fenestration (ISF) could represent an alternative in the treatment of aorto-iliac disease when usual techniques are not available. The aim of this study was to present the results of ISF in aorto-iliac disease. Data will retrospectively be analyzed. Inclusion criteria will be: a surgical abdominal aortic aneurysm (AAA) with an unsuitable anatomy for a standard endograft, aorto-iliac occlusion with narrow distal aorta (<14mm). Technically, after placement of the endograft, a transjugular intrahepatic access set was used to perform ISF. The hole was secondary enlarged using a cutting or non-compliant balloon. Finally, a kissing stent was performed to the aorto- uni-iliac into a bifurcated endograft.

DETAILED DESCRIPTION:
ISF are mainly described at the level of the aortic arch. Different means are reported to perforate the graft: the mechanical (needles, transjugular intra hepatic access needles or guidewires) or physical (laser and radiofrequency catheters).

ISF could be an alternative in the endovascular treatment of aorto iliac disease including both occlusive and aneurysmal pathologies. In this cases, when a narrow distal aorta is present conventional technique as CERAB, bifurcated endograft are challenging. In situ fenestrations allows conversion of an aorto-uni-iliac endograft into a bifurcated endograft, thereby avoiding crossover femorofemoral bypass and its complications.

The aim of the study was to report the results of ISF technique at the level of the abdominal aorta.

Inclusion criteria will be: a surgical abdominal aortic aneurysm (AAA) with an unsuitable anatomy for a standard endograft, aorto-iliac occlusion with narrow distal aorta (<14mm).

All patients had a preoperative CT scan to assess the anatomy of the abdominal aorta.

All patients received an oral antiplatelet agent(aspirin(75-250md/dl) or clopidogrel (75md/dl) and a statin before the procedure.

In situ fenestration technique The procedure was performed under general anesthesia and guided with a mobile C-arm (Siemens). The less diseased and tortuous iliac axis was used to introduce the endograft and the contralateral side as used for the in situ fenestration.

Whenever possible, the procedure was carried out percutaneously with the preclosure technique using Proglide vascular devices for the two common femoral artery retrograde punctures.

The first step consisted in placing an endograft from a retrograde femoral access. The endograft was deployed in a standard fashion. The distal security wire was not released to maintain the control on the distal part of the endograft and keep the graft straight while performing the fenestration. A transjugular intrahepatic access needle was introduced in a 9F Flexor introducer through a contralateral femoral access. When the top of the introducer was at the level of the aortic bifurcation, the dilatator of the introducer was removed, and the introducer was pushed up to the endograft. Contact between the introducer and the endograft was ensured by observing a slight deformation of the endograft while pushing the introducer.

The needle was advanced and the endograft is punctured at the level of the aortic bifurcation. The hole created was secondary enlarged using cutting or high pressure balloon. A long sheath is advanced intro the fenestration to control the success of the technique.

A kissing stent using balloon expandable covered stents is finally performed to stabilize the repair.

Control angiography confirm the patency of the stents and the absence of early endoleak in case of endovascular treatment of abdominal aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

- Underwent in situ fenestration treatment between 2014 and 2019

Exclusion Criteria:

* Patient aged < 40 years or > 90 years
* Under guardianship

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients have been operated with in situ fenestration between 2014 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Primary Patency | at 1 month
  Evaluate primary patency at 1 month after in situ fenestration by CT angiography.
Primary Patency | at 1 month
  Evaluate primary patency at 1 month after in situ fenestration by doppler ultrasound.

SECONDARY OUTCOMES:
Secondary Patency | at 6 and 12 month
  Evaluate secondary patency at 6 and 12 month after in situ fenestration by CT angiography.
Secondary Patency | at 6 and 12 month
  Evaluate secondary patency at 6 and 12 month after in situ fenestration by doppler ultrasound.
Technical success | at baseline
  Technical success was achieved when the perforation of the endograft was performed with the needle. Technical success will be measured as a ratio between the number of successfull perforation and the number of attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël COSCAS, MD, PhD, Principal Investigator — Service de Chirurgie Vasculaire, Hôpital Ambroise Paré; Jérémie JAYET, MD, Study Director — Service de Chirurgie Vasculaire, Hôpital Ambroise Paré
Locations (1):
- Service de Chirurgie Vasculaire, Hôpital Ambroise Paré, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No